CLINICAL TRIAL: NCT01953562
Title: Evaluation of the Influence of Positioning and Time Duration on the Spontaneous Breathing Test in Neonates
Brief Title: Positioning and the Spontaneous Breathing Test in Neonates
Status: Withdrawn | Type: Observational
Why Stopped: This protocol was closed and will be redesigned and submitted as a new protocol.
Sponsor: Christiana Care Health Services (Other)
Responsible Party: Principal Investigator, Robert Locke, Neonatologist, Christiana Care Health Services
Other Study IDs: CCC#33186
Record Dates: First submitted 2013-09-24; First posted 2013-10-01 (Estimated); Last update posted 2016-08-09 (Estimated); Status verified 2016-08

CONDITIONS: Spontaneous Breathing Test; Infants; NICU
Keywords: infants; NICU; intubated; ventilator

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Intubated infants

SUMMARY:
The spontaneous breathing test (SBT) is routinely performed on all intubated patients in the NICU who are potential candidates for extubation from mechanical ventilatory support. For all parents who consent, the routine SBT will be performed on all infants. In addition to the routine SBT the following will occur:

1. work of breathing indices: obtained non-invasively through respiratory inductive plethysmography (RIP).
2. Performing the SBT in the prone position, in addition to the routine position (supine).

ELIGIBILITY:
Inclusion Criteria:

* Infants who qualify for SBT as part of their normal care

Exclusion Criteria:

* Previous history of abdominal or chest surgery (i.e. chest tube, PDA ligation, surgical NEC)
* Congenital malformation of the chest of abdomen
* Neuromuscular disorder
* Current medications affecting neuromuscular tone (ex morphine)
* Unable to be positioned either prone or supine as determined by the attending neonatologist.

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Intubated infants who qualify for the routine spontaneous breathing test.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2013-10; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Effect of prone vs supine positioning on whether an infant receives a passing score on the SBT test | 30 minutes
  SBT is a pass/fail test. The effect of prone vs supine positioning in intubated neonates on whether a spontaneous breathing test is scored pass or fail will be determined.

SECONDARY OUTCOMES:
WOB indices during SBT | 10 minutes
  Determination whether prone vs supine position alters the work of breathing indices in infants while receiving a SBT

CONTACTS AND LOCATIONS:
Overall Officials: Robert Locke, DO, MPH, Principal Investigator — Christiana Care Health Services